CLINICAL TRIAL: NCT00639639
Title: Anti-Tumor Immunotherapy Targeted Against Cytomegalovirus in Patients With Newly-Diagnosed Glioblastoma Multiforme During Recovery From Therapeutic Temozolomide-induced Lymphopenia
Brief Title: Vaccine Therapy in Treating Patients With Newly Diagnosed Glioblastoma Multiforme
Acronym: ATTAC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gary Archer Ph.D. (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Gary Archer Ph.D., Assistant Professor Neurosurgery, Duke University
Organization: Duke University (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00003877; CDR0000589624 (Other: National Cancer Institute); DUMC-8108-07-1R1 (Other: Legacy Duke IRB number); Discretionary Funds (Other: DUMC)
Record Dates: First submitted 2008-03-19; First posted 2008-03-20 (Estimated); Last update posted 2023-03-13 (Actual); Status verified 2023-03

CONDITIONS: Malignant Neoplasms of Brain
Keywords: adult giant cell glioblastoma; adult gliosarcoma
MeSH Terms: conditions — Glioblastoma; Gliosarcoma | interventions — Tetanus Toxoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Arm I (first randomization) (Experimental): Patients receive CMV-ALT IV over 45-90 minutes (course 1 only) and CMV pp65-LAMP mRNA-loaded DC (CMV-DC) vaccine intradermally and administered in equal portions to each inguinal region. Vaccination repeats every 1-3 weeks for up to 3 doses in the absence of unacceptable toxicity.
  Interventions: Biological: therapeutic autologous dendritic cells; Biological: therapeutic autologous lymphocytes
- Arm II (first randomization) (Experimental): Patients receive CMV-DC vaccine intradermally and administered in equal portions to each inguinal region. Vaccination repeats every 1-3 weeks for up to 3 doses in the absence of unacceptable toxicity.
  Interventions: Biological: therapeutic autologous dendritic cells
- Arm I (second randomization) (Experimental): Within 6 to 24 hours prior to vaccination, patients undergo skin site preparation with unpulsed DCs at the vaccination site in one inguinal region. Patients then receive indium In 111-labeled CMV-DC.
  Interventions: Biological: therapeutic autologous dendritic cells
- Arm II (second randomization) (Experimental): Within 6 to 24 hours prior to vaccination, patients undergo vaccination skin site preparation in the opposite inguinal region with tetanus toxoid. Patients then receive 111 In-labeled CMV-DC.
  Interventions: Biological: tetanus toxoid; Biological: therapeutic autologous dendritic cells

INTERVENTIONS:
Biological: tetanus toxoid — Given by injection
  Arms: Arm II (second randomization)
Biological: therapeutic autologous dendritic cells — Given intradermally
Biological: therapeutic autologous lymphocytes — Given IV
  Arms: Arm I (first randomization)

SUMMARY:
RATIONALE: Vaccines may help the body build an effective immune response to kill cancer cells. Radiation therapy uses high-energy x-rays to kill cancer cells. Drugs used in chemotherapy, such as temozolomide, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving vaccine therapy together with radiation therapy and chemotherapy may kill more cancer cells.

PURPOSE: This randomized phase I/II trial is studying how well vaccine therapy works in treating patients with newly diagnosed glioblastoma multiforme recovering from lymphopenia caused by temozolomide.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To evaluate the feasibility and safety of vaccination with cytomegalovirus (CMV) pp65-lysosomal-associated membrane protein (LAMP) mRNA-loaded dendritic cells (DCs) during recovery from therapeutic temozolomide-induced lymphopenia with or without autologous lymphocyte transfer (ALT) in patients with newly diagnosed glioblastoma multiforme and who are seropositive or seronegative for CMV.

Secondary

* To assess humoral and cellular immune responses in these patients to CMV pp65-LAMP mRNA-loaded dendritic cell (CMV-DC) vaccine and to compare the impact of ALT and CMV seropositivity on these parameters.
* To determine if vaccination with or without ALT extends total time to progression or overall survival of these patients when compared to a recent historical cohort.
* To assess the differential ability of indium In^111-labeled DCs to track to the inguinal lymph nodes under different skin preparative conditions.
* To assess the differential ability of ^111In-labeled DCs to track to lymph nodes on the tumor-bearing and non-tumor-bearing side of the cervical lymph nodes.
* To characterize immunologic cell infiltrate in recurrent tumors and seek evidence of antigen escape in recurrent or progressive tumors.

Patients undergo leukapheresis no more than 4 weeks after surgical resection to obtain peripheral blood lymphocytes (PBLs) for human cytomegalovirus (CMV)-autologous lymphocyte transfer (ALT) and CMV-dendritic cell (DC) generation.

Beginning 2-6 weeks after resection, patients undergo external beam radiotherapy (RT) once daily, 5 days a week, for up to 7 weeks. Beginning on day 1 of RT, patients receive oral temozolomide (TMZ) once daily for up to 49 days. Patients with progressive disease during RT, dependence on steroids above physiologic levels, intolerance to TMZ, or failure to meet cell release criteria for DCs or PBLs are removed from study.

Beginning within 2-4 weeks after completion of concurrent RT and TMZ, patients resume oral TMZ once daily on days 1-5. Treatment repeats every 4-6 weeks for up to 6 courses* in the absence of disease progression or unacceptable toxicity. Beginning on day 19-23 of course 1, patients also receive an intradermal immunization. Patients are stratified by CMV serology status (positive vs negative) and are randomized to 1 of 2 vaccine treatment arms.

Note: *Patients may receive additional TMZ treatment at the discretion of the patient and their treating neuro-oncologist.

* Arm I (DC vaccination plus ALT): Patients receive CMV-ALT IV over 45-90 minutes (course 1 only) and 2 x 10^7 CMV pp65-LAMP mRNA-loaded DC (CMV-DC) vaccine intradermally and administered in equal portions to each inguinal region. Vaccination repeats every 1-3 weeks for up to 3 doses in the absence of unacceptable toxicity.
* Arm II (DC vaccination alone): Patients receive CMV-DC vaccine as in arm I. At approximately 2-6 weeks after the third vaccination, all patients undergo a second leukapheresis to obtain peripheral blood mononuclear cells for immunologic monitoring and additional DCs for continued vaccinations. Patients may undergo an additional leukapheresis if they achieve a positive immunological response to therapy or if they require additional DCs to be generated due to a prolonged progression-free survival. Leukapheresis may be performed monthly, but will likely be performed every 4 months throughout the study to generate enough DCs to continue monthly vaccinations.
* Additional cohort (GM-CSF): Patients receive CMV-DC vaccine as in arm II, except that they will also receive GM-CSF in each vaccine. Vaccines continue for a total of 10 unless tumor progression occurs. Patients in this cohort may be enrolled at any point prior to completion of adjuvant TMZ provided they meet all other eligibility criteria.

Prior to the fourth vaccination, patients in both arms and patients with disease progression determined prior to the first scheduled vaccination are stratified according to side of inguinal injection (left vs right) and vaccination skin site preparation (unpulsed DCs vs tetanus toxoid). Patients are then randomized to 1 of 2 treatment arms.

* Arm I (unpulsed DCs): Within 6 to 24 hours prior to vaccination, patients undergo skin site preparation with 1 x 10^6 unpulsed DCs at the vaccination site in one inguinal region. Patients then receive indium In^111-labeled CMV-DC.
* Arm II (tetanus toxoid): Within 6 to 24 hours prior to vaccination, patients undergo vaccination skin site preparation in the opposite inguinal region with tetanus toxoid. Patients then receive indium In^111-labeled CMV-DC as in arm I.

At the time of progression, patients receive a final intradermal vaccination comprising ^111In-labeled CMV-DCs at the base of the jaw bilaterally and to the inguinal region, as a control. Gamma camera images are then taken at 24 and 48 hours after the vaccination to compare DC migration in the groin to each side of the neck injection sites and to observe migration from the neck injection sites to the deep and superficial cervical lymph nodes.

After completion of TMZ therapy, patients continue receiving DC vaccinations in the absence of disease progression (except GM-CSF cohort - total of 10 vaccinations).

Patients undergo blood sample collection periodically for immunologic studies. Samples are examined for functional CD4 and CD8 immune response of patients by cytokine fluorescent cytometry; enumeration of pp65 antigen-specific CD8+ T cells by tetramer analysis; antigen-induced T-cell proliferation; cytokine secretion and quantitative anti-pp65 antibody concentration in the serum by ELISA; and CMV pp65 quantitation in genomic DNA by reverse transcriptase-polymerase chain reaction. Patients may also undergo stereotactic biopsy or tumor resection to confirm tumor progression histologically and to assess immunologic cell infiltration and pp65 antigen escape at the tumor site by immunohistochemistry and polymerase chain reaction.

Quality of life is assessed by the self-reported Functional Assessment of Cancer Therapy-Brain questionnaire at initial leukapheresis, at the first vaccination, after the third vaccination at the time of post-vaccine leukapheresis, and then with every even-numbered vaccination thereafter. A neuropsychological assessment is also conducted prior to the first vaccine and then with every second vaccination thereafter in order to monitor for any changes in neurocognitive or affective changes.

After completion of study therapy, patients are followed periodically.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years of age.
* World Health Organization (WHO) Grade IV glioma with definitive resection prior to leukapheresis with residual radiographic contrast enhancement on most recent CT or MRI of <1 cm in maximal diameter in any axial plane.
* Karnofsky Performance Status (KPS ) of > 80% and a Curran Group status of I-IV.

Exclusion Criteria:

* Radiographic or cytologic evidence of leptomeningeal or multicentric disease at the time of enrollment.
* Prior conventional anti-tumor therapy other than steroids, RT, Avastin or TMZ.
* Pregnant or need to breast feed during the study period (Negative Beta-Human Chorionic Gonadotrophin [HCG] test required).
* Requirement for continuous corticosteroids above physiologic levels at time of first vaccination.
* Active infection requiring treatment or an unexplained febrile (> 101.5o F) illness.
* Known immunosuppressive disease or human immunodeficiency virus infection.
* Patients with unstable or severe intercurrent medical conditions such as severe heart or lung disease.
* Allergic or unable to tolerate TMZ for reasons other than lymphopenia.
* Patients with previous inguinal lymph node dissection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2006-02-06 (Actual); Primary Completion 2017-04-15 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Feasibility and safety of vaccination with cytomegalovirus pp65-LAMP mRNA-loaded dendritic cells (DCs) with or without autologous lymphocyte transfer | 26 months

SECONDARY OUTCOMES:
Humoral and cellular immune responses | 26 months
Time to progression | From time of surgery/diagnosis to date of progression.
Differential ability of indium In-111-labeled DCs to track to the inguinal lymph nodes under different skin preparative conditions | At vaccine # 4
Differential ability of indium In-111-labeled DCs to track to lymph nodes on the tumor bearing and non-tumor bearing side of the cervical lymph nodes | At vaccine # 4
Immunologic cell infiltrate in recurrent tumors | At progression
Evidence of antigen-escape outgrowth in recurrent or progressive tumors | At progression

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Peters, MD, PhD, Principal Investigator — Duke Univeristy Medical Center
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Result] Mitchell DA, Batich KA, Gunn MD, Huang MN, Sanchez-Perez L, Nair SK, Congdon KL, Reap EA, Archer GE, Desjardins A, Friedman AH, Friedman HS, Herndon JE 2nd, Coan A, McLendon RE, Reardon DA, Vredenburgh JJ, Bigner DD, Sampson JH. Tetanus toxoid and CCL3 improve dendritic cell vaccines in mice and glioblastoma patients. Nature. 2015 Mar 19;519(7543):366-9. doi: 10.1038/nature14320. Epub 2015 Mar 11. PMID 25762141
- [Result] Batich KA, Reap EA, Archer GE, Sanchez-Perez L, Nair SK, Schmittling RJ, Norberg P, Xie W, Herndon JE 2nd, Healy P, McLendon RE, Friedman AH, Friedman HS, Bigner D, Vlahovic G, Mitchell DA, Sampson JH. Long-term Survival in Glioblastoma with Cytomegalovirus pp65-Targeted Vaccination. Clin Cancer Res. 2017 Apr 15;23(8):1898-1909. doi: 10.1158/1078-0432.CCR-16-2057. PMID 28411277